CLINICAL TRIAL: NCT01042587
Title: Effect of Bright Light Treatment On Elders In A Long Term Care Environment
Acronym: BrightLights
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Noel H Ballentine, MD, Penn State Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 32704
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-03

CONDITIONS: Behavioral Responses to Bright Light Therapy in Elders
Keywords: bright light therapy; circadian rhythm,; entrainment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bright light (Active Comparator): Bright light has been shown to entrain circadian rhythm so our treatment arm will use thirty minutes of early morning exposure to bright blue light for a four week period.
  Interventions: Other: exposure to bright light
- red light (Sham Comparator): Low level red light is a weak entrainment stimulus of circadian rhythm. Elders in the control group will be exposed to low level red light as a placebo for thirty minutes daily for four weeks.
  Interventions: Other: low luminosity red light

INTERVENTIONS:
Other: exposure to bright light — Elders will be engaged in an activity period which will focus their attention in the direction of bright light, thus ensuring viewing the light source for a daily exposure of thirty minutes.
  Other Names: modified commercially available Phillips Color Graze.
  Arms: bright light
Other: low luminosity red light — Low level red light should not entrain circadian rhythm and will serve as a placebo control
  Other Names: modified commercially available Phillips Color Graze
  Arms: red light

SUMMARY:
The investigators hypothesize that significant exposure to artificial morning bright light (approximately 200 lux of primarily blue light at eye level for thirty minutes daily) as compared to sham bright red light (placebo) will:

1. improve sleep quality
2. improve cognitive scores
3. improve depression scores
4. improve quality of life scores.

DETAILED DESCRIPTION:
Bright light therapy has been shown to improve depression and insomnia in multiple studies. These are common conditions among elders, particularly those residing in long term care environments. Bright light therapy has been inadequately studied in the geriatric population. We will show that a groups of twenty elders can simultaneous be exposed to bright light and that it will result in improvements in multiple realms of behavior and quality of life. Elders will be tested with a number of neuropsychological test batteries prior to exposure to bright light and again at the end of a four week exposure. Some subjects will have daytime and night time activity levels monitored with actigraphy. Cortisol and melatonin levels will be obtained prior to and at the end of the exposure period.

ELIGIBILITY:
Inclusion Criteria:

* residents in Masonic Villages, Elizabethtown, PA long term care
* ability to give informed consent and complete the neuropsychological tests

Exclusion Criteria:

* blindness
* severe illness expected to preclude the ability to complete treatment
* moderate to severe dementia that precludes the ability to complete testing
* light sensitivity making treatment to light therapy uncomfortable

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
assessment of cognitive functioning using MicroCog | once prior to intervention, once near the end of intervention, once four weeks after intervention
Assessment of mood using the Geriatric Depression Scale | once prior to intervention, once near the end of intervention, once four weeks after intervention
assessment of quality of life using the SF-36 | once prior to intervention, once near the end of intervention, once four weeks after intervention
assessment of sleep quality using the Pittsburgh Sleep Quality Index | once prior to intervention, once near the end of intervention, once four weeks after intervention
assessment of mood using the Profile of Moods Survey | weekly throughout the duration of the study
assessment of sleep quality using the Epworth Sleepiness Scale | weekly throughout the duration of the study
day and nightime activity level (5 subjects per group only) using Actigraphy | two weeks prior to light exposure and the second two weeks during light exposure (continuous measurements)

SECONDARY OUTCOMES:
salivary melatonin levels | once prior and near the end of light exposure period
salivary cortisol levels | once prior and near the end of light exposure period

CONTACTS AND LOCATIONS:
Overall Officials: Noel H Ballentine, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Masonic Villages, Elizabethtown, Pennsylvania, United States